CLINICAL TRIAL: NCT04221984
Title: Wingspan One Year Vascular Imaging Events and Neurologic Outcomes (WOVEN)
Brief Title: Wingspan One Year Vascular Imaging Events and Neurologic Outcomes
Acronym: WOVEN
Status: Completed | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Michael J. Alexander, MD, Professor and Vice Chairman, Department of Neurosurgery, Director of the Cedars-Sinai Neurovascular Center, Co-Director, Comprehensive Stroke Center, Cedars-Sinai Medical Center
Other Study IDs: STUDY00000379
Record Dates: First submitted 2020-01-04; First posted 2020-01-09 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Intracranial Atherosclerotic Disease (ICAD)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to determine the one-year post stenting outcomes in patients who were treated with the Wingspan stent on-label in the WEAVE trial. This includes both the assessment of any stroke, hemorrhage, or death, as well as assessment of delayed imaging results to determine the re-stenosis rate of the stents in these patients.

DETAILED DESCRIPTION:
The current study is a retrospective chart and imaging review of the 152 patients enrolled in the WEAVE trial to determine the one-year outcomes for these patients.

This includes both the assessment of any stroke, hemorrhage, or death, as well as assessment of delayed imaging results to determine the re-stenosis rate of the stents in these patients and the medication regimen in those patients who had symptomatic re-stenosis.

The subjects for this study are pre-defined as the 152 patients who had placement of a Wingspan stent for treatment of their intracranial artery stenosis that had symptoms of stroke and 70% or greater arterial stenosis. The study will be conducted at 24 sites in the United States. It is expected that up to 152 patients' records will be assessed for follow up data analysis. Patient's information will be included in the study if they were enrolled in the WEAVE Trial and had placement of a Wingspan stent in its on-label usage indication between 12/1/2013 and 10/31/2017. Follow up information from the patients' charts will be extracted out to the one-year interval following stenting up to December 2018.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for this study are the 152 patients stented in the WEAVE trial on-label.

The patients had the following inclusion criteria:

* Age 18-80
* Intracranial artery stenosis greater or equal to 70% stenosis
* Target artery 2 mm or larger
* Presented with stroke while on medical therapy for stroke prevention
* Prior stroke in the target territory
* Modified Rankin Score of 3 or better (neurologic function)
* Treated greater than 7 days after their last stroke
* Treated with the Wingspan stent by an approved trial NeuroInterventionalist

Exclusion Criteria:

* Patients treated outside of the trial or who did not meet the entry criteria.
* Patients that had stent treatment for arterial dissection
* Patients that had extra-cranial stenosis
* Patients outside the age range of the study
* Patients treated less than 8 days from their stroke.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 152 patients stented on-label in the WEAVE trial.
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2020-05-19 (Actual); Study Completion 2020-05-19 (Actual)

PRIMARY OUTCOMES:
1-year stroke rate following placement of Wingspan stent in this patient cohort | 1 year
  1-year stroke rate following placement of Wingspan stent in this patient cohort
1-year death rate following placement of Wingspan stent in this patient cohort | 1 year
  1-year death rate following placement of Wingspan stent in this patient cohort

SECONDARY OUTCOMES:
Symptomatic re-stenosis rates of the patient group. | 1 year
  Symptomatic re-stenosis rates of the patient group.
Severity of the strokes/index event that occurred in that patient group. | 1 year
  Severity of the strokes/index event that occurred in that patient group.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Alexander, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alexander MJ, Zauner A, Chaloupka JC, Baxter B, Callison RC, Gupta R, Song SS, Yu W; WEAVE Trial Sites and Interventionalists. WEAVE Trial: Final Results in 152 On-Label Patients. Stroke. 2019 Apr;50(4):889-894. doi: 10.1161/STROKEAHA.118.023996. PMID 31125298
- [Background] Bose A, Hartmann M, Henkes H, Liu HM, Teng MM, Szikora I, Berlis A, Reul J, Yu SC, Forsting M, Lui M, Lim W, Sit SP. A novel, self-expanding, nitinol stent in medically refractory intracranial atherosclerotic stenoses: the Wingspan study. Stroke. 2007 May;38(5):1531-7. doi: 10.1161/STROKEAHA.106.477711. Epub 2007 Mar 29. PMID 17395864
- [Background] Chimowitz MI, Lynn MJ, Derdeyn CP, Turan TN, Fiorella D, Lane BF, Janis LS, Lutsep HL, Barnwell SL, Waters MF, Hoh BL, Hourihane JM, Levy EI, Alexandrov AV, Harrigan MR, Chiu D, Klucznik RP, Clark JM, McDougall CG, Johnson MD, Pride GL Jr, Torbey MT, Zaidat OO, Rumboldt Z, Cloft HJ; SAMMPRIS Trial Investigators. Stenting versus aggressive medical therapy for intracranial arterial stenosis. N Engl J Med. 2011 Sep 15;365(11):993-1003. doi: 10.1056/NEJMoa1105335. Epub 2011 Sep 7. PMID 21899409